CLINICAL TRIAL: NCT06198348
Title: Effects of Aerobic Training With and Without Resistance Training on Waist to Hip Ratio, Quality of Life and Menstrual Dysfunction in Polycystic Ovarian Syndrome.
Brief Title: Aerobic Training With and Without Resistance Training in Polycystic Ovarian Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S22C14G92023
Record Dates: First submitted 2023-12-26; First posted 2024-01-10 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Polycystic ovarian syndrome; Quality of life; Waist to Hip Ratio; Aerobic Exercise; Resistance Training
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Exercise; Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic Exercise (Control Group) (Other): Group A will receive Aerobic exercise plan. The treatment will be given with the frequency of 3 times per week for 8 weeks. Treatment sessions will be of 30 minutes with short resting intervals
  Interventions: Other: Aerobic Exercise
- Aerobic exercise with resistance training (Experimental Group) (Experimental): Group B will receive aerobic and resistance exercise plan. The frequency of treatment will be as same as that of aerobic exercise program i.e. 3 times a week for 8 weeks. Treatment sessions will be of 45 minutes with short resting intervals
  Interventions: Other: Aerobic Exercises with Resistance training

INTERVENTIONS:
Other: Aerobic Exercise — Treatment Protocol to Group A It consists of patients who will receive aerobic exercise sessions 3 times per week for 8 weeks. Every session will be of 30 minutes.
  It will include warm up phase, active phase and cool down phase Warm-up phase:
  In which each participant will walk at 80 m/min at for 5 min.
  Active phase:
  Brisk walking or treadmill:
  In which each participant will perform brisk walking for 15 mints initially. After that gradually duration of brisk walking will increase.
  Arms: Aerobic Exercise (Control Group)
Other: Aerobic Exercises with Resistance training — These groups will perform these exercises:
  Aerobic exercise +resistance exercises Exercise
  Session: 3 days per week Time of exercise session: 30-45 min
  After following protocol of aerobic exercise as mentioned above the subjects will perform resistance exercises. These Exercises will perform:
  1. Leg press (dual leg press):
     Leg press targets the Glutes "Quadriceps or quads .but they also work your "Hamstrings".
  2. Crunches:
     Crunches Target the abdominal muscles specifically rectus abdominis and obliques.
  3. Squats:
  Squats targets the adductor muscles of the hip, glutes and rectus abdominis muscle Leg Extension
  Total Exercise plan for 12 weeks:
  1-2 weeks: Repitations: 10-15 times
  No of sets: 1 set Resistance: minimum 3-4 weeks:
  Repitations: 10-15 times
  No of sets: 2 set Resistance: moderate 5-6 weeks:
  Repitations: 15-16 times
  No of sets: 2 set Resistance: moderate 7-8 weeks:
  Repitations: 15-16 times No of sets: 2 set
  Arms: Aerobic exercise with resistance training (Experimental Group)

SUMMARY:
Polycystic ovary syndrome (PCOS) characterized by a chronic disorder in ovulation along with hyperandrogenism has become one of the most common endocrine disorders in women of reproductive age with an estimated 5%-15% prevalence. It has the symptoms such as menstrual disorders, infertility, hyperandrogenism, obesity, hirsutism and acne. PCOS is linked to Psychological morbidities e.g. increased risk of stress, depression, low self-esteem, poor body image, and reduced health-related quality of life. Approximately 75% of people with PCOS have a fat accumulation in the central area of the body.

DETAILED DESCRIPTION:
A Randomized controlled trial will be conducted to determine the effects of Aerobic training with and without resistance training on the waist to hip ratio, QoL and menstrual dysfunction in polycystic ovarian syndrome. A sample size of 22 PCOS women's will be taken, Data will be collected from Jinnah Hospital Lahore by using PCOSQ and SF-36 questionnaire. A written consent form will be taken from participants meeting inclusion criteria and will be randomly allocated into two groups of equal members. One group undergoing aerobic with resistance exercise training i.e., the experimental group and other with aerobic exercise i.e., control group. The interventions will be provided for 30 mints for 3 days per week for 2 months. All participants in both groups will be evaluated before and after the treatment programs.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40yrs
* Waist to hip ratio >87(20)
* Women who are diagnosed according to Rotterdam criteria e.g. oligo/anovulation, hyperandrogenism, and polycystic ovaries.(21)
* Female who physically able to performs exercise

Exclusion Criteria:

* Women who are smoking and using drugs for depression.
* Married women
* Women with other pathological conditions like diabetes and thyroid diseases.
* Females who are not able to perform resistant exercise

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Polycystic Ovary Syndrome only occurs in females.
Enrollment: 22 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
SF-36 Questionnaire | 8 weeks
  QoL was assessed by the validated Portuguese version of the self-reported MOS SF-36, which consists of eight subscales: (1) Physical Role Function, (2) Physical Functioning, (3) Bodily Pain, (4) General Health Perception, (5) Vitality, (6) Social Role Functioning, (7) Emotional Role functioning, and (8) Mental Health. A substantial body of research supports the reliability of the SF-36 measurements.validity of SF-36 Questionnaire is 0.90 Subscale scores range from 0 to 100, with a lower score indicating lower QoL for that subscale.
Self-administered PCOSQ | 8 weeks
  All the participants filled up the self-administered PCOSQ. PCOS Questionnaire has 26 items divided into 5 domains: emotions (8 items), body hair (5 items), weight (5 items), infertility (4 items), and menstrual problems (4 items). Each question is associated with a 7point scale in which 7 represents optimal function and 1 represents the poorest Function. PCOSQ dimensions were internally reliable with Cronbach's a scores ranging from 0.70 to 0.97.
Measuring Tape | 8 weeks
  Waist circumference (WC) was measured with the participant in the standing position, with arms at the side of the body, feet together, and with a relaxed abdomen. For WC, a horizontal measurement was obtained on the narrower part of the dorsum (above the navel and below the xiphoid process.
  Hip circumference (HC) was measured using the same positioning, as the region with the largest circumference of the buttocks. Waist-to-hip ratio (WHR) was measured by dividing the WC value by the HC value

CONTACTS AND LOCATIONS:
Overall Officials: Faiza Taufiq, PPDPT, Principal Investigator — Riphah International University, Senior Lecturer
Locations (1):
- Jinnah Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No